CLINICAL TRIAL: NCT03321864
Title: Capture of Prostatic Trans-rectal Ultrasound Scans for Research Into Improved Targeted Biopsy Techniques (CAPTURE)
Brief Title: Capture of Prostatic Trans-rectal Ultrasound Scans for Research
Acronym: CAPTURE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left Trust currently.
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, David Thurtle, Clinical Research Associate and Honorary Urology Registrar, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A094516; 228575 (Registry Identifier: IRAS ID)
Record Dates: First submitted 2017-10-13; First posted 2017-10-26 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer; Prostate Neoplasm
Keywords: Transperineal biopsy; Prostate cancer; Transrectal ultrasound; Fusion biopsy techniques
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: All available patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): All patients recruited to the study (this arm) will have an additional transrectal ultrasound whilst already under GA for TP biopsy.
  Interventions: Procedure: Transrectal ultrasound scan of prostate

INTERVENTIONS:
Procedure: Transrectal ultrasound scan of prostate — Additional transrectal ultrasound whilst already under GA for transperineal biopsy.

SUMMARY:
Through this study the investigators seek to build up a repository of prostate ultrasonography videos and prostate MRI scans to enable research into novel anatomical registration techniques. These data will facilitate the development of improved technology that enables targeting of tumours seen on MRI using free-hand biopsy techniques, without the need for a gantry or overlaid perineal grid.

DETAILED DESCRIPTION:
The purpose of this study is to explore whether mathematical and computational modelling techniques can be used to enable anatomical based real-time image registration for guiding prostate biopsies. This would lead to the ability to perform free-hand trans-perineal biopsy without the need for supporting gantries or a biopsy grid placed over the perineum. This will significantly decrease costs of trans-perineal biopsy, reduce the number of puncture sites through the perineal skin - reducing pain and bleeding - and reduce the procedure time. Alongside locally developed local-anaesthetic transperineal biopsy techniques it will allow targeted biopsy to be taken in the outpatient setting, improving patient convenience, and helping health services to meet growing demands on targeted biopsies.

The investigators aim to create a new method of mapping the prostate using free-hand ultrasound, without any additional physical equipment. This may require collaborations with approved International groups with particular skills in relevant mathematical or engineering techniques.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing trans-perineal prostate biopsy under general anaesthesia who have had an MRI of their prostate within the preceding 12 months.
* Male.
* Age 18-100.

Exclusion Criteria:

* Those unable to provide informed consent.
* Any medical condition, vital sign or laboratory value that, in the opinion of the investigator or responsible anaesthetist makes any prolongation of general anaesthesia unsafe to the participant.
* Patients unable to have an MRI

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Prostate size | Years 1-5
  Ultrasound images and videos of the prostate will be captured to measure the length, width and depth of the prostate on ultrasound. The measurements will be in millimeters (mm). This will be taken at a single time-point at the time of general anaesthesia for transperineal biopsy.
Prostate location | Years 1-5
  Ultrasound images and videos of the prostate will be captured to assess prostate location relative to surrounding structures. Specifically this will mean measuring the distance from the anal verge to the prostate. Unit of measurment is millimeters (mm). This will be taken at a single time-point at the time of general anaesthesia for transperineal biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: David Thurtle, Principal Investigator — University of Cambridge
Locations (1):
- Addenbrookes Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No